CLINICAL TRIAL: NCT00148889
Title: Prospective,Randomised, Double-blind, Multicenter Study to Assess the Efficacy and Safety of Bilateral Globus Pallidus Internus - in Patients With Medically Refractory Primary Cervical Dystonia
Brief Title: Double-blind, Multicenter Study to Assess the Efficacy of Bilateral Pallidal Stimulation in Patients With Medically Refractory Primary Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German Parkinson Study Group (GPS) (Other)
Collaborators: Medtronic (Industry); Competence Network on Parkinson's Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD-DBS-2005-JM
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cervical Dystonia
Keywords: cervical dystonia; torticollis; deep brain stimulation; pallidal stimulation; globus pallidus internus
MeSH Terms: conditions — Torticollis | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Sham Comparator): Sham-stimulation
  Interventions: Device: Deep brain stimulation (DBS)
- 1 (Active Comparator): Active GPI-DBS
  Interventions: Device: Deep brain stimulation (DBS)

INTERVENTIONS:
Device: Deep brain stimulation (DBS) — Bilateral pallidal stimulation with an implanted DBS device

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of bilateral pallidal stimulation in patients with medically refractory primary cervical dystonia.

DETAILED DESCRIPTION:
Primary cervical dystonia (CD) affects about 20-40/100.000 population. The disease is chronic and life-long. The therapy of choice are local intramuscular Botulinum Toxin injections given every three months. Oral medication such as anticholinergics or dopamine depleting drugs are usually of limited efficacy or their use is limited by intolerable side-effects. About 5-10% of CD patients develop neutralizing antibodies against Botulinum Toxin. Two previous controlled multicenter trials have shown the efficacy and safety of bilateral pallidal stimulation in patients with primary segmental and generalized dystonia (one study was performed by our group).

Following surgery, patients will be randomized 1:1 to verum or placebo stimulation for a period of three months. Primary outcome measure is the TWSTRS (Toronto Western Spasmodic Torticollis Rating Scale) - a validated and widely accepted physician-based outcome measure for cervical dystonia. The independent TWSTRS raters are movement disorders specialists unaware of the stimulation status (verum/placebo) and they compare the TWSTRS-score at baseline and 3-months follow-up. Our hypothesis is that stimulated patients will have a significantly better improvement of dystonia as compared to those without stimulation (placebo group).

After the 3-months period, all patients are unblinded and receive continuous effective stimulation by the implanted system. Regular follow-up visits are scheduled every 12 months for 5 years postoperatively to assess the long-term efficacy of pallidal stimulation. Side-effects are assessed in a standardized way and include the assessment of surgery-induced as well as stimulation-induced side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Primary cervical dystonia
* Disease duration 3 years or longer
* Adult patient (18 years or older)
* TWSTRS severity score 15 or more
* Non-response to Botulinum Toxin
* Non-response to oral antidystonic medication
* Informed consent

Exclusion Criteria:

* Dementia (Mattis Dementia Rating Scale below 120)
* Severe depression (Beck Depression Inventory >25)
* Previous functional stereotactic surgery
* Hemidystonia or generalized dystonia
* Severe brain atrophy
* Contraindication against surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Scale (TWSTRS) at 3 months following surgery (comparison between placebo and control group) | 3 months

SECONDARY OUTCOMES:
side-effects, quality of life, depression, pain, long-term efficacy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Mueller, MD, Principal Investigator — Department of Neurology, Medical University Innsbruck, Anichstr. 35, A-6020 Innsbruck, Austria
Locations (10):
- Austria (2):
  - Medical University Innsbruck, Department of Neurology, Innsbruck, Tyrol
  - Department of Neurosurgery, Medical University Vienna, Vienna
- Germany (8):
  - Department of Neurology, Charité, Humboldt-University Berlin, Berlin
  - Department for Stereotaxy and Functional Neurosurgery, University Cologne, Cologne
  - Clinic of Neurosurgery, Medical University Hannover, Hanover
  - Department of Neurology, University Heidelberg, Heidelberg
  - Department of Neurology, University Kiel, Kiel
  - Department of Neurology, University Regensburg, Regensburg
  - Department of Neurology, University Rostock, Rostock
  - Hertie-Institute for Clinical Brain Research, Tübingen

REFERENCES:
- [Derived] Dinkelbach L, Mueller J, Poewe W, Delazer M, Elben S, Wolters A, Karner E, Wittstock M, Benecke R, Schnitzler A, Volkmann J, Sudmeyer M. Cognitive outcome of pallidal deep brain stimulation for primary cervical dystonia: One year follow up results of a prospective multicenter trial. Parkinsonism Relat Disord. 2015 Aug;21(8):976-80. doi: 10.1016/j.parkreldis.2015.06.002. Epub 2015 Jun 4. PMID 26074391
- [Derived] Volkmann J, Mueller J, Deuschl G, Kuhn AA, Krauss JK, Poewe W, Timmermann L, Falk D, Kupsch A, Kivi A, Schneider GH, Schnitzler A, Sudmeyer M, Voges J, Wolters A, Wittstock M, Muller JU, Hering S, Eisner W, Vesper J, Prokop T, Pinsker M, Schrader C, Kloss M, Kiening K, Boetzel K, Mehrkens J, Skogseid IM, Ramm-Pettersen J, Kemmler G, Bhatia KP, Vitek JL, Benecke R; DBS study group for dystonia. Pallidal neurostimulation in patients with medication-refractory cervical dystonia: a randomised, sham-controlled trial. Lancet Neurol. 2014 Sep;13(9):875-84. doi: 10.1016/S1474-4422(14)70143-7. Epub 2014 Aug 7. PMID 25127231
- See also: Homepage Competence Network on Parkinson's disease sponsored by the German government — http://www.kompetenznetz-parkinson.de